CLINICAL TRIAL: NCT04338568
Title: Accuracy and Inter-observer Variability of Lung Ultrasound in COVID-19 Pneumonia
Brief Title: Screening COVID-19 by Point-of-care Lung Ultrasound: a Validation Study
Acronym: SCOUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Prof. dr. Michiel Thomeer, Prof.Dr.Michiel Thomeer, Hasselt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTU2020032
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: COVID-19 Pneumonia; Lung Ultrasound
Keywords: accuracy; inter-observer variability

STUDY DESIGN:
Intervention Model Description: Patients with the diagnosis of COVID-19 pneumonia will undergo a lung ultrasound, by two observers each. The findings will be compared with findings on chest x-ray and/or CT thorax. Accuracy and inter-observer variability will be calculated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS observer 1 (Active Comparator): The subject will undergo a Lung Ultrasound by observer nr 1
  Interventions: Diagnostic Test: Lung ultrasound
- LUS observer 2 (Active Comparator): The subject will undergo a Lung Ultrasound by observer nr 2
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — The lung ultrasound examination consists of two-sided scanning of the anterior and lateral chest wall and is performed with patients in supine or near-to-supine position.

SUMMARY:
COVID-19 is a rapidly spreading and very contagious disease caused by a novel coronavirus that can lead to respiratory insufficiency. In many patients, the chest radiograph at first presentation be normal, and early low-dose CT-scan is advocated to diagnose viral pneumonia. Lung ultrasound (LUS) has similar diagnostic properties as CT for diagnosing pneumonia. However, it has the advantage that it can be performed at point-of-care, minimizing the need to transfer the patient, reducing the number of health care personnel and equipment that come in contact with the patient and thus potentially decrease the risk of spreading the infection.

This study has the objective to examine the accuracy of lung ultrasound in patients with proven COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. high probability CT thorax or chest X-ray for viral pneumonia within five days of the day of inclusion
2. positive COVID-19 nasopharyngeal swab within 10 days of inclusion
3. 18 years or older
4. Oxygen saturation of < 93% in ambient air
5. Signed written informed consent

Exclusion Criteria:

* Contra-indication for lung ultrasound
* Other causes of hypoxia or of pulmonary infiltrates on CT thorax or chest X-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the diagnosis of interstitial syndrome by lung ultrasound | within 2 weeks after first subject included
  The diagnostic accuracy of lung ultrasound is more than 90% compared to low-dose CT or chest X-ray for the detection of viral pneumonia in patients with COVID-19 infection.
Inter-observer variability | within 2 weeks after first subject included
  The interobserver variability by lung ultrasound between the 2 observers for the diagnosis of interstitial syndrome by lung ultrasound is > 0.6 measured by the Kappa score

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Thomeer, MD,PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Background] Ramirez P, Torres A. Should ultrasound be included in the initial assessment of respiratory patients? Lancet Respir Med. 2014 Aug;2(8):599-600. doi: 10.1016/S2213-2600(14)70142-0. Epub 2014 Jul 3. No abstract available. PMID 24998675
- [Result] Pisani L, Vercesi V, van Tongeren PSI, Lagrand WK, Leopold SJ, Huson MAM, Henwood PC, Walden A, Smit MR, Riviello ED, Pelosi P, Dondorp AM, Schultz MJ; Lung Ultrasound Consortium. The diagnostic accuracy for ARDS of global versus regional lung ultrasound scores - a post hoc analysis of an observational study in invasively ventilated ICU patients. Intensive Care Med Exp. 2019 Jul 25;7(Suppl 1):44. doi: 10.1186/s40635-019-0241-6. PMID 31346914
- [Result] Li K, Fang Y, Li W, Pan C, Qin P, Zhong Y, Liu X, Huang M, Liao Y, Li S. CT image visual quantitative evaluation and clinical classification of coronavirus disease (COVID-19). Eur Radiol. 2020 Aug;30(8):4407-4416. doi: 10.1007/s00330-020-06817-6. Epub 2020 Mar 25. PMID 32215691
- Available data/document: Clinical Study Report — https://www.castoredc.com/